CLINICAL TRIAL: NCT03327142
Title: EUS-guided FNA in the Study of the Adrenal Gland: National Retrospective Multicenter Study
Brief Title: EUS-guided FNA in the Study of the Adrenal Gland
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, JOAN B GORNALS, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: AdrenalG EUS-Study
Record Dates: First submitted 2017-03-29; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-08

CONDITIONS: Adrenal Gland Disease; Adrenal Tumor
Keywords: Adrenal Gland; Endoscopic Ultrasound Guided FNA
MeSH Terms: conditions — Adrenal Gland Diseases; Adrenal Gland Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopic Ultrasound-Guided FNA — Endoscopic Ultrasound Guided Fine Needle Aspiration of Puncture of Adrenal Glands
  Other Names: Endosonography

SUMMARY:
To analyze the diagnostic performance, safety, impact on clinical management, predictors of malignancy and cyto-pathological correlation of the EUS-FNA with AG. National multicenter retrospective study. Mailing-SEED partners. Participation: 17 Spanish centers. Inclusion period: April / 2003 to April / 2016 Inclusion criteria: All AG (Left / Right) punctured by EUS.

A review of 205 EUS-FNA of AG in 200 patients is included.

DETAILED DESCRIPTION:
INTRODUCTION: The EUS has proven useful in the study and evaluation of the adrenal gland (AG) by endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA), in both the left and right glands.

OBJECTIVE: To analyze the diagnostic performance, safety, impact on clinical management, predictors of malignancy and cyto-pathological correlation of the EUS-FNA with AG.

MATERIALS AND METHODS: National multicenter retrospective study. Mailing-SEED partners. Participation: 17 Spanish centers. Inclusion period: April / 2003 to April / 2016 Inclusion criteria: All AG (Left / Right) punctured by EUS. Variables reviewed: Demographic characteristics, clinical, extension studies, USE and pathological data. Comparison between variables; and estimation of multivariate logistic model for cytology, mortality and therapeutic change.

ELIGIBILITY:
Inclusion Criteria:

* All adrenal gland (Left / Right) punctured by endoscopic ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nationwide. Mailing-invitation to Spanish Society of Digestive Endoscopy (SEED) partners. Participation: 17 Spanish centers.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | retrospective analysis form 2003 to 2016

SECONDARY OUTCOMES:
number of adverse events related to the procedure | retrospective analysis, last 10 years
Predictors of malignancy | retrospective analysis, last 10 years
  Predictors of malignancy and cyto-pathological correlation of the EUS-FNA with adrenal gland

IPD SHARING:
Plan to Share IPD: Undecided